CLINICAL TRIAL: NCT06698185
Title: A Clinical Phase II Study of the Materna Device to Shorten Delivery Time During Childbirth
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in IRB jurisdiction for study, study is suspended
Sponsor: Materna Medical (Industry)
Collaborators: El Camino Hospital, Mountain View, CA (Unknown); Altos Oaks Medical Group, Mountain View, CA (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MAT-2002
Record Dates: First submitted 2016-03-14; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Childbirth
Keywords: Childbirth, Tearing, perineal lacerations, pelvic muscle, avulsion, pelvic floor disorders, vaginal delivery, instrument delivery, delivery time, ultrasound
MeSH Terms: conditions — Lacerations; Fractures, Avulsion; Pelvic Floor Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Materna Prep Device (Experimental): Materna Prep Device
  Interventions: Device: Materna Prep Device
- Sham Control (Sham Comparator): Sham Control
  Interventions: Device: Sham Control

INTERVENTIONS:
Device: Materna Prep Device — Materna Prep Device
  Arms: Materna Prep Device
Device: Sham Control — Sham Control
  Arms: Sham Control

SUMMARY:
This feasibility study is a prospective, non-randomized, single arm study to evaluate safety and prevention of maternal pelvic soft-tissue damage using the Materna Medical Device. The device will be used during the first stage of labor, following initiation of epidural anesthesia and after the cervix has dilated to between 3-8 cm. Up to 20 subjects will be included in the initial study, with the option to increase the number of subjects to 50 based on early data.

DETAILED DESCRIPTION:
Study Inclusion Criteria are:

1. Patients attending for antenatal care at El Camino Hospital with the Altos Oaks Obstetrics Group
2. First ongoing pregnancy beyond 20 weeks
3. Singleton, cephalic presentation
4. No pregnancy complications which are likely to require Caesarean Section
5. Planned vaginal delivery

The primary outcome measure is device safety as defined by freedom of device related adverse events. Secondary efficacy outcome measures are:

1. Pelvic muscle damage as determined by ultrasound imaging
2. Length of the 2nd stage of labour
3. Delivery mode
4. Perineal and anal sphincter trauma
5. Symptoms of incontinence, prolapse and sexual dysfunction 2 years postpartum
6. Pelvic organ support (ICS POP-Q system) and pelvic organ descent on ultrasound

Interested patients will have the study presented to them during their pre-natal visits with the Altos Oaks Obstetrics group. Interested patients will have the study explained to them and will be given the Informed Consent document.After the informed consent procedure, patients will undergo an interview and 4D translabial ultrasound.

The screened patients will have the Materna device administered by a researcher from the Altos Oaks Obstetrics group. The patients will be flagged in their charts regarding their participation in this study. When an enrolled patient arrives at the hospital and is deemed to be in labor, the Altos Oaks physician on call will be notified, and called to administer the use of the device. All other obstetric services are provided by routine staff. The device will be dilated up to a maximum diameter of 8-10cm and is then removed to allow delivery. The Control arm patients will experience normal care during labor. Participants are followed up at 3 months and 1 year after childbirth with an interview, including validated questionnaires on bladder, bowel and sexual function, and repeat ultrasound. Delivery details will be collected by the midwives and through the institutional database.

The study's primary efficacy outcome measure is levator avulsion injury diagnosed on volume ultrasound data obtained at the 1-3 month follow-up appointment. Secondary outcomes include both objective findings related to pelvic floor function and anatomy, as well as symptoms of pelvic floor dysfunction such as pelvic organ prolapse, urinary / fecal incontinence and dyspareunia, as ascertained by interview and questionnaire, at 3 months after childbirth. Assessment of stored ultrasound volume data (obtained on pelvic floor muscle contraction, or, if that is not possible, at rest) is undertaken at a later date by one single operator within the Altos Oaks Obstetrics group.

ELIGIBILITY:
Inclusion Criteria:

1. Primiparas, or previous pregnancy terminated before 24 weeks gestation
2. Single fetus birth
3. Subject is able to understand the risks and potential benefits of participating in the study and is willing to provide written informed consent.
4. Subject is willing and able to comply with specified follow-up evaluations.
5. Planned to have epidural during birthing process

Exclusion Criteria:

1. Previous delivery, or previous pregnancy beyond 24 weeks gestation
2. Less than 36 weeks gestation
3. Neurological diseases e.g. Multiple Sclerosis that may result in unrelated pelvic disorders
4. Muscular or skin disorder that affects elasticity of tissue such as scleroderma or lupus.
5. Local or systemic infection e.g. HIV, herpes
6. Any prior surgical procedures to the vaginal anatomy that could lead to pelvic dysfunction, pelvic fractures, or pelvic soft tissue injuries. Evaluated during baseline screening
7. High likelihood of less than 1 hour of potential device dilation time after the woman arrives at the center and receives epidural

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Safety | 3 months post-delivery follow-up
  Freedom from device related adverse events

SECONDARY OUTCOMES:
Pelvic Muscle Avulsion | 1-3 months post delivery
  Binary, determined with ultrasound imaging
Pelvic Muscle Damage | 1-3 Months Post-Delivery
  Measured by changes in levator hiatus area, determined with ultrasound imaging
Delivery Time | Immediate after delivery
  Measure the length of the second phase of labor
Perineal Lacerations | Immediate Post Delivery
  Record the grade of perineal lacerations, and if sutures were used to repair lacerations
Instrument Deliveries | Immediate Post-Delivery
  Record if instruments were used for delivery

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Weber, MD, Principal Investigator — Obstatrician, Altos Oaks Medical Group
Locations (1):
- El Camino Hospital, Mountain View, California, United States